CLINICAL TRIAL: NCT04967677
Title: Establishing of the Inter-rater Reliability and Variability of Selected Standardized Tests Performed According to New Czech Extended Manuals
Brief Title: Establishing of the Inter-rater Reliability and Variability of Selected Standardized Tests Performed in Czech Language
Status: Active, not recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Rybářová, Mgr. Kateřina Rybářová (Master in Occupational Therapy), Charles University, Czech Republic
Other Study IDs: 96/20 Grant GA UK 2. LF UK
Record Dates: First submitted 2021-05-30; First posted 2021-07-19 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Motor Activity
Keywords: standardized test; occupational therapy; fine motor skills; Nine Hole Peg Test; Purdue Pegboard Test; Box and Block Test; inter-rater reliability; variability; Czech language
MeSH Terms: conditions — Motor Activity | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Czech healthy occupational therapy students: Czech healthy occupational therapy students will be asked to fill in a questionnaire. Then they will be tested by the Nine Hole Peg Test, the Purdue Pegboard Test and the Box and Block Test. Video of their performance will be obtained.
  Interventions: Diagnostic Test: Nine Hole Peg Test, Purdue Pegboard Test, Box and Block Test

INTERVENTIONS:
Diagnostic Test: Nine Hole Peg Test, Purdue Pegboard Test, Box and Block Test — At first, each person will be asked to fill in the questionnaire. Than he/she will be tested by the Nine Hole Peg Test, Purdue Pegboard Test and the Box and Block Test according to the Czech version of extended manuals for those tests. Audio recording of verbal instructions will be used.
  Other Names: questionnaire

SUMMARY:
The main aim of the pilot project is to establish inter-rater reliability, internal variability and variability of results got in two different ways of the Nine Hole Peg Test, Purdue Pegboard Test and Box and Block Test administered according to the new Czech extended versions of their manuals.

DETAILED DESCRIPTION:
New Czech manuals for the Nine Hole Peg Test, Purdue Pegboard Test and Box and Block Test were made by back-translation method. They were updated and extended by new rules for unification of their performing. The manuals include instructions for performing three trials of each subtest.

At least 30 occupational therapy students will be tested by those three tests according to those new Czech manuals. Video of students' performance will be obtained.

The inter-rater reliability, internal variability and variability of results got in two different ways will be established.

ELIGIBILITY:
Inclusion Criteria:

* Czech language as a mother tongue
* age from 20 to 65 years
* occupational therapy student

Exclusion Criteria:

* diagnosed pathology of the upper limbs or diseases that negatively affect the dexterity of their limbs
* use of drugs affecting attention
* vision impairment uncorrectable with glasses
* severe hearing loss
* inability to understand instructions
* inability to read or write
* inability to complete complete testing
* failure to sign Informed consent for probation with inclusion to research and Consent to the collection and processing of personal data during the study at the General University Hospital in Prague

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-representation
Study Population: Czech healty occupational therapy students
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
results from the Nine Hole Peg Test | 10 minutes
  time in seconds and hundredth of seconds
results from the Purdue Pegboard Test | 25 minutes
  number of parts put in the Pegboard according to the rules
results from the Box and Block Test | 30 minutes
  number of transported blocks

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Rybářová, Mgr., Principal Investigator — Charles University And General University Hospital In Prague
Locations (1):
- Department of Rehabilitation Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No